CLINICAL TRIAL: NCT06672029
Title: Long-term Effectiveness of Integrative Scoliosis-specific Rehabilitation in High-risk Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin-Fen Hsieh, Study Principal Investigator, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20241003R
Record Dates: First submitted 2024-10-24; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: adolescent idiopathic scoliosis; manual therapy; Schroth Best Practice; Gensingen brace; scoliosis-specific rehabilitation program

STUDY DESIGN:
Intervention Model Description: retrospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with adolescent idiopathic scoliosis (Experimental): All patients receive a combination of therapy including the three listed below:
  * The pattern-specific manual therapy
  * The Schroth Best Practice exercises
  * The Gensingen brace application
  Interventions: Other: combining pattern-specific manual therapy, Schroth Best Practice exercise, and Gensingen brace application

INTERVENTIONS:
Other: combining pattern-specific manual therapy, Schroth Best Practice exercise, and Gensingen brace application — * The pattern-specific manual therapy: It was developed by our author. This therapy was done immediately before each SBP (Schroth Best Practice) exercise session, targeting both the spine and extra-spinal regions.
  * The Schroth Best Practice exercises: It contains following 6 components: The physio-logic® program for sagittal profile correction, education on activities of daily living (ADLs), the "3D made easy" program, the new "Power Schroth" program, the rehabilitation of walk, and neuromobilization.
  * The Gensingen brace application: it was made according to the patients' Lehnert Schroth Classifications. the investigators recommended the patients to wear the brace for 21-23 hours per day during the first year. As the bone maturation reached Risser 4 to 4.5, the daily brace wearing time was gradually reduced.

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is one of the most common spinal deformities diagnosed in adolescents, especially female, with the prevalence in general population ranging from 0.93% to 12%, 80% of which are idiopathic. The management and treatment of AIS includes observation, physiotherapy (or therapeutic exercise), brace application, and surgery. Evidence of the conservative management of AIS has been stronger in recent years. However, the best combination therapy has not been well established. Moreover, the investigator has demonstrated an innovation of pattern-specific manual therapy to treat AIS. Different from previous conservative treatment, the investigators applied specific treatment for different patterns of AIS according to the Lehnert-Schroth (LS) scoliosis classification. Therefore, the investigators aim to determinate the long-term effects of the integrative scoliosis-specific rehabilitation program combining pattern-specific manual therapy, Schroth Best Practice (SBP) exercise, and Gensingen brace application in treating AIS patients.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is one of the most common spinal deformities diagnosed in adolescents, especially female, with the prevalence in general population ranging from 0.93% to 12%, 80% of which are idiopathic. It is a complex 3D structural disorder, diagnosed when the Cobb angle is equal to or greater than 10 degrees, accompanied by vertebral rotation. The risk factors of curve progression include growth spurt, positive family history, laxity of skin and joints, flat back, and angle of trunk rotation more than 10 degrees. Curve progression can lead to aesthetic concerns, spinal pain syndromes, and respiratory dysfunction.

The management and treatment of AIS includes observation, physiotherapy (or therapeutic exercise), brace application, and surgery. According to Lonstein et al, a progression factor, which is used for the risk assessment of curve progression of progression, is calculated using the Risser sign, age at presentation, and magnitude of the curve. A probability for progression of under 40% is indicated for observation only, while the probability for progression of 40% - 60% is indicated for physiotherapy, and the probability for progression of over 60% is considered indicated for bracing application. Current evidence recommended that bracing be applied in evolutive AIS patients (Risser 0 to 3) with curves above 20° ± 5° Cobb.

Current studies have investigated the efficacy of conservative treatment for AIS. In terms of bracing, previous studies have shown that AIS patients treated with Rigo Chêneau orthoses had lower major curve progression versus those with Boston-style orthoses. Furthermore, the Gensingen brace is developed from Chêneau brace with individual computer-aided design, which exhibits efficacy in decreasing Cobb angle and angle of trunk rotation. There are a wide range of physiotherapeutic scoliosis-specific exercise methods, among which the Schroth exercise program is the mostly studied and is proven to be effective. The Schroth method consists of postural, sensorimotor, and corrective breathing exercises in daily activities for three-dimensional correction of the patients' specific curve patterns.

A randomized-controlled study in 2016 revealed that Schroth exercise program was superior to home exercise and control groups in decreasing the Cobb and rotation angles. In addition, a randomized-controlled study in 2016 revealed that adding Schroth physiotherapeutic scoliosis-specific exercises to standard care of bracing can lead to better reduction of curve severity than bracing alone in treating AIS patients. Also, long-term improvement of combining Schroth exercise and Chêneau orthoses has been observed. On the other hand, manual therapy in treating AIS is less studied, and current evidence is insufficient to confirm the benefit of manual therapy in AIS patients. This study applied a pattern-specific manual therapy to mobilize and realign the asymmetry of the spine and extra-spinal regions.

Evidence of the conservative management of AIS has been stronger in recent years. However, the best combination therapy has not been well established. Moreover, the investigator has demonstrated an innovation of pattern-specific manual therapy, to treat AIS. Different from previous conservative treatment, the investigators applied specific treatment for different patterns of AIS according to the Lehnert-Schroth (LS) scoliosis classification. Therefore, the investigators aim to determinate the long-term effects of the integrative scoliosis-specific rehabilitation program combining pattern-specific manual therapy, Schroth Best Practice exercise, and Gensingen brace application in treating AIS patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) fulfill a diagnosis of AIS;
* 2) age between 10 and 18 years old;
* 3) Cobb angle ≧ 20˚;
* 4) incidence of progression over 60% according to Lonstein et al. ;
* 5) never underwent treatment that might affect scoliosis;
* 6) complete follow-ups of at least 12 months after the end of treatment.

Exclusion Criteria:

* 1) A diagnosis of non-idiopathic scoliosis (e.g. secondary or functional scoliosis);
* 2) any psychological problems;
* 3) pregnancy;
* 4) any severe rheumatic or chronic neuromuscular diseases (e.g. rheumatoid arthritis, ankylosing spondylitis);
* 5) any severe orthopedic problems (e.g. bone tumor, fracture);
* 6) refusal of the suggested treatment;
* 7) any previous or ongoing treatment of scoliosis;
* 8) any contraindications to brace, exercise, or manipulative treatment.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Angle of trunk rotation (ATR) | measured at the baseline, end of the treatment course (about half an year), and a year after the treatment course
  The ATR was measured with a Scoliometer™ in a forward bending posture. It is defined as the angle between the horizontal plane and the plane across the posterior aspect of the back, and the minimal clinically important difference (MCID) is 5 degrees.
Cobb angle | measured at the baseline, end of the treatment course (about half an year), and a year after the treatment course
  The Cobb angles of major curves were measured via standing posteroanterior radiograph. Based on the consensus of SOSORT and SRS non-operative management committee, radiographic definitions of improvement is 6 degrees or more.

SECONDARY OUTCOMES:
lateral deviation | measured at the baseline, end of the treatment course (about half an year), and a year after the treatment course
  Lateral deviation, which may affect trunk balance, is measured by the distance between transitional point (TP) and central sacral line via posteroanterior whole spine radiograph. It was measured only for those with TP deviation more than 2 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, M.D., Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan